CLINICAL TRIAL: NCT04784481
Title: Ivermectin Reproposing for COVID-19 Treatment in Outpatients With Mild Stage
Brief Title: Ivermectin Reproposing for Mild Stage COVID-19 Outpatients
Acronym: IVER-Leve
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ministry of Public Health, Argentina (Other Government)
Responsible Party: Principal Investigator, Maria de los Angeles Peral de Bruno, Director of Research - Ministry of Health of Tucumán, Ministry of Public Health, Argentina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5077-410-CH2020
Record Dates: First submitted 2021-02-20; First posted 2021-03-05 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome)
Keywords: Ivermectin; Outpatient; Mild stage; Health Primary Center
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Cluster-randomised trials.
Masking Description: Each of the health centers (cluster of health centers) was randomly assigned to receive or not the intervention under study. The conglomerate of outpatients randomly assigned to the Experimental Group (EG) and Control Group (CG) belongs to the urban and peri-urban areas from Tucumán, and the selection of the centers was carried out considering a homogeneous socioeconomic profile in relation to the operating areas in which it is organized the Public Health Systems. Participants were recruited prior to cluster randomisation. Staff of each assistance center knew what intervention was being implemented as well as patients. Data processing group was blind to analyze the database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The EG received Ivermectin orally 4 tablets of 6 mg = 24 mg every 7 days for 4 weeks.
  All participants were evaluated by physical examination COVID-19 diagnosed with positive RT-PCR at the beginning, and final of the protocol
  Interventions: Drug: Ivermectin
- Control Group (No Intervention): Conventional treatment. All participants were evaluated by physical examination COVID-19 diagnosed with positive RT-PCR at the beginning, and final of the protocol

INTERVENTIONS:
Drug: Ivermectin — Experimental Group received Ivermectin orally 4 tablets of 6 mg = 24 mg every 7 days for 4 weeks.
  Other Names: N/D
  Arms: Experimental Group

SUMMARY:
Background:

The emergency of COVID-19, along with the current difficulties in responding to the high demand for vaccines, requests to the scientific community to find alternative treatments based on reuse of drugs as a strategy to prevent the progression of the disease in patients infected with SARS COV 2.

Objetive This study aims to evaluate the use of ivermectin in mild-stage patients to increase outpatient discharge and prevent the progression to moderate or severe stages of the disease.

Added value of this study We found that an intervention with ivermectin has impacted on the PPS in a population of outpatients care, between the 5th and 9th day. Also, the treatment increased the probability to obtain outpatient discharge, even in the presence of comorbidities.

Implications of all available evidence.

Research in Context According to the COVID-19 Treatment Guidelines by the NIH, most trials have several limitations. It needs results from adequately powered and well-designed clinical trials to provide evidence-based guidance on the role of ivermectin in the treatment of COVID- 19. However, our study shows overlaps in benefits with other authors, and taking together, these results are encouraging for further study about repurposing ivermectin for the treatment of COVID-19.

DETAILED DESCRIPTION:
Technical Design:

Cluster Randomised Trials in outpatients care, n = 254. The subjects were divided into experimental (EG: n = 110) and control groups (CG: n = 144). The criteria for this choice were based on the geographical distribution of Health Services, locomotion, and logistics in current times of pandemic.

Sample Size:

Sample size was determined by the test comparing two proportions. It considered the following parameters to the bilateral test: n = 30,000 Total operating area population for services network to Primary Care; 95% confidence level, 3% precision, 5% proportion, n = 201 sample size without loss, 20% expected proportion of losses. The sample size calculated was n= 252 participants.

Participants:

The total group n = 254 enrolled outpatients care from the urban area-department heads and peri-urban area of the City San Miguel de Tucumán. The study was conducted between September 2020 to January 2021. The health coverage service was administered by the Health System of the State of Tucumán (SI.PRO.SA, Tucumán, Argentina). The people who agreed to participate in the study gave their informed consent before starting the study (Research Ethics Committee / Health Research Directorate, file number 054/2020).

Intervention Protocol:

The EG received protocol ivermectin orally 4 tablets of 6 mg = 24 mg every 7 days for 4 weeks plus symptomatic treatment (500mg paracetamol every 6 or 8h, no more than 4 tablets daily;100mg aspirin, 1 tablet per day with breakfast; 150mg Ranitidine, 1 tablet in the morning, and 1 tablet at night). The CG received only symptomatic treatment. Patients with comorbidities continued with the basic medication for the underlying pathology . All participants were evaluated by physical examination and COVID-19 infection was diagnosed with positive RT-PCR. Clinical evaluation of symptoms was carried throughout the study period. Enrolled subjects completed symptom questionnaires (including reporting of any adverse effects of treatment), physical examinations and remote clinical telemedicine follow-up and received outpatient discharge 4 weeks after the start of the intervention.

The 10-category ordinal scale recommended by the WHO was used to classify patients according to clinical patient state: ambulatory mild disease, moderate disease, severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients infected by SARSCoV-2 confirmed either by RT-PCR test, Neo Kit or rapid test authorized by ANMAT or by close contact or epidemiological link;
* Women of childbearing age with a negative pregnancy test;
* Mild disease-patients with two or more of the following symptoms: fever less than 38·5°C and higher than 37.5°C according to Ministry of Health, Argentina(16), isolated diarrheal episodes, hyposmia or hypogeusia, mild desaturation (between 96 and 93%), dyspnea, polyarthralgia, persistent headache, abdominal pain, erythema of the kidney, nonspecific rash.

Exclusion Criteria:

* Hypersensitivity or allergy to Ivermectin;
* Pregnant or lactating;
* Children or adolescents under 18 years of age;
* Patients with Neurological Pathology, Renal Insufficiency, Hepatic Insufficiency;
* Weight less than 40kg;
* Patients with concomitant use of drugs that act on GABA, barbiturate and benzodiazepine receptors;
* Patients who have not completed / signed the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Proportion test | from 5th to 9th day.
  a) Proportion of patients with symptoms (fever, diarrhea, taste and/or smell disturbance, SpO2, polyarthralgia, headache, body pain, abdominal pain, ALRI symptoms and signs)
Proportion test | from 10th to 14th day.
  Proportion of patientts with symptoms (fever, diarrhea, taste and/or smell disturbance, SpO2, polyarthralgia, headache, body pain, abdominal pain, ALRI symptoms and signs)

SECONDARY OUTCOMES:
Odd Ratio | 28 days after enrollment
  Medical release: numbers of participants with absence of clinical symptoms relation to COVID-19 disease.
Odd Ratio and logistic regression test | 28 days after enrollment
  Relative risk of being cured "with" or "without" treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rossana E. Chahla, MD. Ph.D., Principal Investigator — Ministery of Health, Tucumán, Argentina
Locations (1):
- SI.PRO.SA, Ministerio de Salud Pública, San Miguel de Tucumán, Argentina

IPD SHARING:
Plan to Share IPD: No
N/D

REFERENCES:
- [Background] Bacchetti P, Leung JM. Sample size calculations in clinical research. Anesthesiology. 2002 Oct;97(4):1028-9; author reply 1029-32. doi: 10.1097/00000542-200210000-00050. No abstract available. PMID 12357184
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Ashburn TT, Thor KB. Drug repositioning: identifying and developing new uses for existing drugs. Nat Rev Drug Discov. 2004 Aug;3(8):673-83. doi: 10.1038/nrd1468. No abstract available. PMID 15286734
- [Background] Liu Z, Fang H, Reagan K, Xu X, Mendrick DL, Slikker W Jr, Tong W. In silico drug repositioning: what we need to know. Drug Discov Today. 2013 Feb;18(3-4):110-5. doi: 10.1016/j.drudis.2012.08.005. Epub 2012 Aug 28. PMID 22935104
- [Background] Gonzalez Canga A, Sahagun Prieto AM, Diez Liebana MJ, Fernandez Martinez N, Sierra Vega M, Garcia Vieitez JJ. The pharmacokinetics and interactions of ivermectin in humans--a mini-review. AAPS J. 2008;10(1):42-6. doi: 10.1208/s12248-007-9000-9. Epub 2008 Jan 25. PMID 18446504
- [Result] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768